CLINICAL TRIAL: NCT00392392
Title: Phase II Study of Preoperative Bevacizumab and Trastuzumab Administered With ABI-007 and Carboplatin in HER2 Overexpressing Breast Cancer
Brief Title: Preoperative Bevacizumab and Trastuzumab With ABI-007 and Carboplatin in HER2+ Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI BRE 83
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2013-02-13 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Bevacizumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients received treatment with nab-paclitaxel (100 mg/m2 IV days 1, 8, 15) and carboplatin (AUC 6 IV day 1) every 28 days for 6 cycles. Trastuzumab (4 mg/kg loading dose, followed by 2 mg/kg) and bevacizumab (5 mg/kg IV) were administered weekly for 23 weeks, beginning concurrently with chemotherapy. Patients then underwent either mastectomy or breast conserving surgery and pathologic treatment responses were assessed. After surgery, trastuzumab 6 mg/kg and bevacizumab 15 mg/kg were administered at 3 week intervals for a total of 52 weeks.
  Interventions: Drug: nab-paclitaxel; Drug: Bevacizumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: nab-paclitaxel — ABI-007
  Other Names: Abraxane; ABI-007
Drug: Bevacizumab — Bevacizumab
  Other Names: Avastin
Drug: Trastuzumab — Trastuzumab
  Other Names: Herceptin

SUMMARY:
This trial combines trastuzumab and bevacizumab monoclonal antibodies, with ABI-007 and carboplatin, as neoadjuvant therapy in previously untreated locally advanced breast cancers demonstrating HER2 gene amplification. It is hoped that this novel combination will result in increased pathologic response rates that will translate into long term outcome improvements in HER2 positive patients with locally advanced breast cancer.

DETAILED DESCRIPTION:
All eligible patients will receive induction chemotherapy prior to consideration of primary surgical intervention. If surgical intervention is deemed not to be in the best interest of the patient, patient will go off study at the time of evaluation for surgery. Upon completion of chemotherapy and surgery, all ER + and/or PR + patients will be placed on Tamoxifen 20 mg/qd or an aromatase inhibitor.

Induction preoperative therapy:

* Bevacizumab
* Trastuzumab
* ABI-007
* Carboplatin

Postoperative Adjuvant Therapy:

* Bevacizumab
* Trastuzumab

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically confirmed adenocarcinoma of the breast or inflammatory breast cancer
* Clinical stage T 1-4, N 0-3, M0
* FISH+ HER2 gene amplified breast cancer
* 18 years or older
* Normal cardiac function
* Performance status 0-2
* Cannot have received any prior chemotherapy for this disease or cannot have received chemotherapy for any other cancer in the past 5 years.
* Previous diagnosis of noninvasive breast cancer is OK.
* Must have adequate bone marrow, renal and liver function.
* Pregnant or lactating females not allowed.
* Preexisting peripheral neuropathy must be equal to or less than grade 1
* Must have archived tumor tissue for tissue testing.

Exclusion Criteria:

You cannot be in this study if you any of the following:

* History of cardiac disease, with New York Heart Association Class II or greater with congestive heart failure
* Any heart attack, stroke or TIAs within the last 6 months or serious arrhythmias needing medication; no bleeding diathesis or coagulopathy.
* No prior investigational drug within the last 30 days
* No prior trastuzumab or bevacizumab therapy

There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Yardley, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Background] Yardley DA, Raefsky E, Castillo R, Lahiry A, Locicero R, Thompson D, Shastry M, Burris HA 3rd, Hainsworth JD. Phase II study of neoadjuvant weekly nab-paclitaxel and carboplatin, with bevacizumab and trastuzumab, as treatment for women with locally advanced HER2+ breast cancer. Clin Breast Cancer. 2011 Oct;11(5):297-305. doi: 10.1016/j.clbc.2011.04.002. Epub 2011 May 5. PMID 21729666

RESULTS

PARTICIPANT FLOW:
Groups:
- Nab-Paclitaxel/Bevacizumab/Trastuzumab: Patients received treatment with nab-paclitaxel (100 mg/m2 IV days 1, 8, 15) and carboplatin (AUC 6 IV day 1) every 28 days for 6 cycles. Trastuzumab (4 mg/kg loading dose, followed by 2 mg/kg) and bevacizumab (5 mg/kg IV) were administered weekly for 23 weeks, beginning concurrently with chemotherapy. Patients then underwent either mastectomy or breast conserving surgery and pathologic treatment responses were assessed. After surgery, trastuzumab 6 mg/kg and bevacizumab 15 mg/kg were administered at 3 week intervals for a total of 52 weeks.
Period: Overall Study
Arm/Group | Nab-Paclitaxel/Bevacizumab/Trastuzumab
Started | 29
Completed | 9
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Nab-Paclitaxel/Bevacizumab/Trastuzumab
Number analyzed (Participants) | 29
Age Continuous [Median (Full Range); unit: years] | 52 [29 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate (PCRR), the Percentage of Patients Who Have No Evidence of Cancer in the Breast or Lymph Nodes Following Surgery
Description: Pathologic complete response was defined as the absence of residual invasive cancer in the breast (pT0) and axillary lymph nodes (pN0).
Time Frame: 18 months
Population: Two patients refused surgery after completing six cycles of pre-operative (neoadjuvant) therapy.
Measure: Number; unit: percentage of participants
Arm/Group | Nab-Paclitaxel/Bevacizumab/Trastuzumab
Number analyzed (Participants) | 27
percentage of participants | 56

ADVERSE EVENTS:
Arm/Group | Nab-Paclitaxel/Bevacizumab/Trastuzumab
Serious Adverse Events (participants affected / at risk) | 8/29
Other Adverse Events (participants affected / at risk) | 29/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-Paclitaxel/Bevacizumab/Trastuzumab (N=29)
Pain - Abdomen (General disorders) | 1 (1)
Infection - Skin (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
Pain - Chest (General disorders) | 1 (1)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 1 (1)
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Infection - Sepsis (Infections and infestations) | 2 (2)
Creatinine (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-Paclitaxel/Bevacizumab/Trastuzumab (N=29)
Alopecia (Skin and subcutaneous tissue disorders) | 19 (77)
ALT (Hepatobiliary disorders) | 7 (17)
Anorexia (Gastrointestinal disorders) | 5 (6)
AST (Hepatobiliary disorders) | 4 (14)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 5 (5) — Decreased LVEF
Rigors/Chills (General disorders) | 2 (3)
CO2 (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 11 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Creatinine (Renal and urinary disorders) | 2 (3)
Mood Alteration - Depression (Psychiatric disorders) | 3 (8)
Diarrhea (Gastrointestinal disorders) | 16 (30)
Dizziness (Nervous system disorders) | 7 (13)
Edema (Blood and lymphatic system disorders) | 3 (3)
Fatigue (General disorders) | 25 (118)
Fever (General disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 29 (184)
Hemorrhage Pulmonary - Nose (Respiratory, thoracic and mediastinal disorders) | 19 (40)
Hemorrhage, GI - Rectal (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GU (Renal and urinary disorders) | 3 (4)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Hot Flashes (Endocrine disorders) | 4 (10)
Allergic Reaction (Immune system disorders) | 2 (2)
Hypertension (Cardiac disorders) | 15 (40)
Infection - Breast (Infections and infestations) | 2 (3)
Infection - Sepsis (Infections and infestations) | 2 (2)
Infection - Sinusitis (Infections and infestations) | 8 (18)
Infection - URI (Infections and infestations) | 3 (4)
Infection - UTI (Infections and infestations) | 4 (5)
Insomnia (General disorders) | 8 (11)
Leukocytes (Blood and lymphatic system disorders) | 26 (109)
Lymphopenia (Blood and lymphatic system disorders) | 2 (15)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (41)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (8)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (5)
Mood Alteration - Anxiety (Psychiatric disorders) | 11 (31)
Mucositis (Gastrointestinal disorders) | 9 (16)
Nausea (Gastrointestinal disorders) | 25 (58)
Neuropathy - NOS (Nervous system disorders) | 4 (15)
Neuropathy - Sensory (Nervous system disorders) | 11 (33)
Neutrophils (Blood and lymphatic system disorders) | 27 (116)
Pain - Abdomen (General disorders) | 3 (4)
Pain - Back (General disorders) | 6 (12)
Pain - Bone (General disorders) | 3 (9)
Pain - Breast (General disorders) | 3 (9)
Pain - Chest (General disorders) | 8 (12)
Pain - Headache (General disorders) | 18 (39)
Pain - Joint (General disorders) | 8 (13)
Pain - Limb (General disorders) | 8 (23)
Pain - Muscle (General disorders) | 8 (9)
Pain - Neck (General disorders) | 3 (5)
Pain - NOS (General disorders) | 3 (4)
Pain - Oral (General disorders) | 4 (6)
Pain - Throat (General disorders) | 3 (6)
Pain - Urinary (General disorders) | 4 (4)
Palpitations (Cardiac disorders) | 2 (4)
Phlebitis (Vascular disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 21 (68)
Proteinuria (Renal and urinary disorders) | 7 (15)
Pruritis (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatitis - Radiation (Skin and subcutaneous tissue disorders) | 4 (6)
Acne (Skin and subcutaneous tissue disorders) | 2 (6)
Rash (Skin and subcutaneous tissue disorders) | 10 (20)
Esophagitis (Gastrointestinal disorders) | 9 (21)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (8)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Sweating (General disorders) | 4 (6)
Tachycardia (Cardiac disorders) | 2 (2)
Taste Alteration (Gastrointestinal disorders) | 7 (19)
Urinary Frequency (Renal and urinary disorders) | 2 (5)
Ocular - Visual Changes (Eye disorders) | 3 (5)
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Vomiting (Gastrointestinal disorders) | 8 (23)
Weakness (General disorders) | 2 (3)
Weight Gain (General disorders) | 2 (2)
Wound Complication (Skin and subcutaneous tissue disorders) | 4 (7)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.